CLINICAL TRIAL: NCT02228798
Title: Perioperative Anticoagulant Use (Dabigatran, Rivaroxaban, or Apixaban) for Elective Surgery/Procedure Evaluation in Patients With Atrial Fibrillation (AF).
Brief Title: Perioperative Anticoagulant Use for Surgery Evaluation Study
Acronym: PAUSE
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, James Douketis, Dr. James Douketis-Principal Investigator, McMaster University
Other Study IDs: CIHR-PAUSE-2014; CIHR313156 HSFG-14-0006163 (Other Grant/Funding Number: CIHR, HSF)
Record Dates: First submitted 2014-08-25; First posted 2014-08-29 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation
Keywords: anticoagulant; atrial fibrillation; surgery; oral anticoagulant; discontinue; DOAC; NOAC; blood thinner; interruption
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (platelet deprived plasma) will be collected on day of surgery/procedure and measured by 'everyday' coagulation tests that are not DOAC-specific (e.g., activated partial thromboplastin time [aPTT]) and 'specialized' coagulation tests that are DOAC-specific (dilute thrombin time [TT] - HemoclotTM, and anti-factor Xa assays) to determine the effect of the pre-operative DOAC interruption protocol on the level of residual anticoagulation.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Rivaroxaban: Patients currently taking rivaroxaban that have atrial fibrillation and require surgery or a procedure.
- Dabigatran: Patients currently taking dabigatran that have atrial fibrillation and require surgery or a procedure.
- Apixaban: Patients currently taking apixaban that have atrial fibrillation and require surgery or a procedure.

SUMMARY:
The aim of the Perioperative Anticoagulant Use for Surgery Evaluation (PAUSE) Study, is to establish a safe, standardized protocol for the perioperative management of patients with atrial fibrillation (AF) who are receiving a novel oral anticoagulant (DOAC) drug, either dabigatran, rivaroxaban or apixaban, and require an elective surgery/procedure.

DETAILED DESCRIPTION:
The primary aim is to demonstrate that a standardized but patient-focused protocol for the perioperative management of each DOAC is safe, with acceptably low rates of perioperative major bleeding (MB) and arterial thromboembolism (ATE). The perioperative protocol is adjusted based on patient renal function and surgery/procedure-related bleed risk, to optimize patient safety, and does not involve heparin bridging anticoagulation.

The secondary aim of the PAUSE Study is to determine the effect of the pre-operative DOAC interruption protocol on the level of residual anticoagulation, when measured by 'everyday' coagulation tests that are not DOAC-specific (e.g., activated partial thromboplastin time [aPTT]) and 'specialized' coagulation tests that are DOAC-specific (dilute thrombin time [TT] - HemoclotTM, and anti-factor Xa assays).

Approximately 3,300 patients from 15 to 25 centres over a 3.5 year period will be recruited across Canada for the PAUSE Study.

Patients with Atrial Fibrillation and are currently taking dabigatran, rivaroxaban and apixaban (DOACs) and require elective surgery/procedure will follow a standardized management perioperative protocol for discontinuation of their DOAC prior to surgery. Patients will be discontinuing the DOAC they are currently receiving from 1 to 4 days prior to surgery or procedure, depending on bleed risk, type of DOAC, and creatinine clearance rate.

A blood sample will be taken on the day of the surgery or procedure for measurement of laboratory outcomes (residual level of anticoagulant on day of surgery).

Patients will be followed up weekly up to a month for primary outcome assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Receiving a DOAC (dabigatran or rivaroxaban or apixaban) for Atrial Fibrillation
3. Ability to assess patient at lease one day prior to DOAC discontinuation

Exclusion Criteria:

1. CrCl less than 30 mL per min for dabigatran- and rivaroxaban-treated patients ( less than 25 mL per min for apixaban-treated patients) as estimated by Cockroft-Gault formula
2. Cognitive impairment or psychiatric illness that precludes collection of followup data
3. Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those patients who are currently taking dabigatran, rivaroxaban or apixaban for oral anticoagulation used for stroke prevention in atrial fibrillation, and who require its temporary interruption for a surgical or other procedure, will be recruited from 15 to 25 participating sites across Canada.
  The study plans to screen 4,114 patients over a 3 year period, with 80 per cent expected enrollment (3,291 patients) from 16 sites across Canada. Equal number of patients, per oral anticoagulant arm will be enrolled, with approximately 1,000 patients taking each DOAC.
Sampling Method: Non-Probability Sample
Enrollment: 3135 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Major Bleeds | Within 30 days of surgery or procedure
  The first primary outcome is Major Bleed:Bleeding that is fatal or is symptomatic and retroperitoneal, intracranial, intraspinal, intraocular, pericardial, intramuscular with compartment syndrome, or intra-articular.
  Non-surgical bleeding causing a drop in hemoglobin greater than or equal to 20 g per L or leading to transfusion greater or equal to 2 units of blood within 24 hours.Surgical bleed that leads to intervention or interferes with mobilization or leads to delayed wound healing; or leads to deep wound infection.
  Surgical site bleeding that is unexpected and prolonged and or sufficiently large to cause hemodynamic instability associated with a drop in hemoglobin greater or equal to 20 g per L or transfusion of greater or equal to 2 units of blood within 24 hours.
  The second primary outcome is atrial thromboembolism (ATE), comprising: Ischemic stroke,Systemic embolism: symptomatic embolism to upper or lower extremity or abdominal organ or transient ischemic attack.
Number of participants with Atrial Thromboembolism | Within 30 days of surgery or procedure
  The second primary outcome is atrial thromboembolism (ATE), comprising:
  * Ischemic stroke: any new focal neurologic deficit that persists for >24 hours or any new focal neurologic deficit of any duration, that occurs with evidence of acute infarction on computed tomography (CT) or magnetic resonance imaging (MRI) of the brain.
  * Systemic embolism: symptomatic embolism to upper or lower extremity or abdominal organ, confirmed intra-operatively or by objective imaging studies (e.g. CT angiography).
  * Transient ischemic attack: symptomatic focal neurologic deficit (lasting typically less than 1 hour), that occurs with no evidence of acute infarction on CT or MRI of brain.

SECONDARY OUTCOMES:
Number of participants with Minor bleeding | 30 days or less after surgery or porcedure
  • Minor bleeding: bleeding not satisfying criteria for major bleeding; investigator will report bleeding events using pertinent clinical data and with an assessment from the surgeon.
Number of participants who die | 30 days or after surgery or procedure
  Death: death due to any cause.
Number of participants that have a Venous Thromboembolism (VTE) | 30 days or less after surgery
  Venous thromboembolism (VTE): comprising symptomatic deep vein thrombosis and pulmonary embolism, confirmed by objective imaging studies (e.g., ultrasound, CT pulmonary angiogram).
Number of participants who acquire Acute Coronary Syndrome | 30 days or less after surgery or procedure
  • Acute coronary syndrome: symptomatic myocardial ischemia, defined by pre-specified clinical and objective EKG- and/or troponin-related criteria N.B. Patients who develop any clinical outcome will be treated according to standards of care.

OTHER OUTCOMES:
Dilute TT test-Laboratory blood test of NOAC levels | Day of Surgery
  • DOAC levels will be measured by the dilute TT test expressed in ng/mL.
Anti-Xa test for NOAC level | Day of surgery
  DOAC levels as measured by an anti-Xa tests, expressed in ng/mL.
INR Laboratory Test | Day of surgery
  • The INR will be done to compare these tests with novel oral anticoagulant specialized Anti-Xa tests
PT Laboratory test | Day of surgery
  PT will be measured to compare these tests with novel oral anticoagulant specialized Anti-Xa tests
aPTT Laboratory test | Day of Surgery
  To compare these tests with novel oral anticoagulant specialized Anti-Xa tests
TT Laboratory test | Day of surgery
  To compare these tests with novel oral anticoagulant specialized Anti-Xa tests

CONTACTS AND LOCATIONS:
Overall Officials: James Douketis, MD, Principal Investigator — McMaster University/St. Joseph's Healthcare
Locations (21):
- United States (3):
  - Department of Pharmacy, Kaiser Permanente Colorado, Aurora, CO, USA, Aurora, Colorado
  - NorthShore University HealthSystem, Evanston, Illinois
  - Henry Ford Health System, Detroit, Michigan
- Department of Cardiovascular Sciences, University of Leuven, Leuven, Belgium
- Canada (15):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - QEII Hospital, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - North York General, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - University of Manitoba, Winnipeg, Ontario
  - Maisonneuve-Rosemont, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Montreal Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital, Montreal, Quebec
- Department of Anesthesiology, University of Thessaly, Larissa, Greece
- Department of Vascular Medicine, Amsterdam Cardiovascular Sciences, Amsterdam, Netherlands

REFERENCES:
- [Derived] Shaw JR, Li N, Vanassche T, Coppens M, Spyropoulos AC, Syed S, Radwi M, Duncan J, Schulman S, Douketis JD. Predictors of preprocedural direct oral anticoagulant levels in patients having an elective surgery or procedure. Blood Adv. 2020 Aug 11;4(15):3520-3527. doi: 10.1182/bloodadvances.2020002335. PMID 32756938